CLINICAL TRIAL: NCT05873738
Title: Smoking Cessation is Associated With Short-term Improvement of Vascular Health in a Cohort of People Living With HIV in Rio de Janeiro, Brazil.
Brief Title: Smoking Cessation in a Cohort HIV+ Rio de Janeiro, Brazil.
Status: Completed | Type: Observational
Sponsor: Instituto Fernandes Figueira (Other Government)
Responsible Party: Principal Investigator, Rodrigo de Carvalho Moreira, Dr, Oswaldo Cruz Foundation
Other Study IDs: 3.171.692
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation; Brachial Flow Mediated Dilatation; Nicotine Replacement Therapy
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Relapse
  Interventions: Drug: Nicotine replacement
- Group 2: Smoking cessation
  Interventions: Drug: Nicotine replacement

INTERVENTIONS:
Drug: Nicotine replacement — Nicotine patches

SUMMARY:
The study was carried out within a large, urban prospective cohort of PLHIV at the Instituto Nacional de Infectologia Evandro Chagas (INI). Located in Rio de Janeiro, Brazil, INI is a national public referral center for PLWHA receiving primary care since 1998. From December 2019, adults who had attitudes toward quitting smoking and had no contraindications to study pharmacotherapy were enrolled by active site searching

ELIGIBILITY:
Inclusion Criteria:

* individuals were deemed as regular smokers, defined as the consumption of one or more pack (20 cigarettes) per week in the past 6 months, and expired carbon monoxide (CO) measurement > 10 ppm at the screening visit.

Exclusion Criteria:

* previous use of transdermal nicotine patches or bupropion in the last 6 months; (ii) contraindication to nicotine patches; (iii). Pregnancy; (iv) breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults HIV positive who had attitudes toward quitting smoking and had no contraindications to study pharmacotherapy
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
FMD | 12 months
  Flow mediated brachial artery dilatation

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Infectologia Evandro Chagas, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
Upon request data will be shared , anonimyzed